CLINICAL TRIAL: NCT05641402
Title: Developing Evidence-based Text Messages to Target Diet and Physical Activity Behaviour for People with Type 2 Diabetes Mellitus
Brief Title: Evidence-based Text Messages to Target Diet and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: University of Oxford (Other); Manchester University NHS Foundation Trust (Other Government); Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Yvonne Kiera Bartlett, Lecturer, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIHR202832
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experienced acceptability study (Other): The final study in this research will involve people with type 2 diabetes receiving the text messages
  Interventions: Other: Text messages

INTERVENTIONS:
Other: Text messages — Text messages based on behaviour change techniques

SUMMARY:
This research aims to develop a bank of text messages based on behaviour change techniques targeting specific diet and physical activity behaviours in people with type 2 diabetes

DETAILED DESCRIPTION:
Aim: To develop text messages that help people with type 2 diabetes (T2D) improve their diet and level of physical activity

What is known:

Following diet and physical activity advice helps to reduce the risk of health problems for people with T2D

Just telling people about a healthy diet, or ideal levels of physical activity may not change what someone does day-to-day. Many people need support to change health behaviours

Techniques designed to help people change their behaviour, such as setting goals, can help people act

Text messages can be sent to large numbers of people, for a low cost

For the best chance of success, it is important that the messages are a) acceptable to the people receiving them and b) use techniques to help people to make changes

How the investigators are going to achieve their aim:

When asking someone to follow a healthy diet or do more physical activity, this could refer to changing lots of different behaviours such as eating less sugar or less fat and walking each day. The investigators invited people with type 2 diabetes, doctors, nurses, dietitians, and researchers to take part in a workshop to work out which behaviours are the most important ones for people with type 2 diabetes to do. The investigators have also looked at previous research and found techniques that have helped people with type 2 diabetes change their diet and levels of activity.

The investigators will now follow four steps to develop the messages:

1. Twelve to fifteen people with type 2 diabetes will take part in online focus groups to provide feedback about the target behaviours and guide the development of the text message system
2. Ten to twenty researchers will take part in a workshop. They will write messages using the techniques that have worked in previous research to target important behaviours for people with type 2 diabetes. They will then complete a survey to report whether the messages are good examples of the techniques.

2. Sixty people with type 2 diabetes will complete a survey to tell us whether they like and understand the messages and how useful they think they would be.

3. Forty people with type 2 diabetes will receive the messages for up to 3 months and take part in an interview over the phone to help us understand their experiences.

Patient and Public Involvement and Engagement (PPIE) This research has been developed with a PPIE group. Our PPIE co-applicant and PPIE group will be involved in key decisions and review any materials being sent to people with type 2 diabetes.

What the investigators will do with the findings

Explore how these messages can become part of routine National Health Service (NHS) care. The findings will be used together with work our team are doing looking at sending out text messages to help people with type 2 diabetes take their medication.

Findings will also be publicised through databases of people interested in research, diabetes charities, community groups, places of worship and publications.

ELIGIBILITY:
* For the expert workshop -

Inclusion criteria: researchers with expertise in behaviour change, physical activity, diet and/or diabetes

- For focus group

Inclusion criteria

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 years or above.
* A diagnosis of type 2 diabetes.
* Has access to a mobile-phone (shared access is allowed with permission of phone owner)
* Able to use a mobile phone, if necessary with help, to send or retrieve brief messages (including text-messages or messaging within smartphone applications).

Exclusion criteria

Moved out of England prior to taking part in the study

For the anticipated acceptability survey and experienced acceptability study

Inclusion criteria

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18 years or above.
* A diagnosis of type 2 diabetes.
* Has access to a mobile-phone (shared access is allowed with permission of phone owner)
* Able to use a mobile phone, if necessary with help, to send or retrieve brief messages (including text-messages).

Exclusion criteria

* Within three months of a hospital admission for hyperglycaemia or hypoglycaemia.
* Pregnant or within three months post-partum by self-report
* Underweight (For anticipated acceptability this will be by self-report, for experienced acceptability BMI<18.5)
* Historical or current diagnosis of an eating disorder Prescribed insulin for their diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Experienced Acceptability of the text messages for people with type 2 diabetes | 3.5 months
  Assessed through interviews following receiving the text messages

SECONDARY OUTCOMES:
Anticipated Acceptability | 60 minutes
  Assessed through online survey
Rating of fidelity to intended behaviour change technique | 60 minutes
  How well the text messages represent their intended behaviour change technique. For each behaviour change technique, participants will be presented with the title and description of the technique from the Behaviour change Technique (BCT) v1 taxonomy (Michie et al., 2013, doi: 10.1007/s12160-013-9486-6), and then sample messages. For each message participants will be asked "How well does this message reflect the [specific technique] as defined above?". Answers were given on a 10-point scale anchored with 1 (not very well) to 10 (very well).
  This scale has been used in our previous work developing text messages (Bartlett et al., 2020, doi: 10.2196/15989)

CONTACTS AND LOCATIONS:
Overall Officials: Kiera Bartlett, PhD, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Subject to participant consent. Plan to upload the deidentified survey data with codebook Will explore uploading deidentified transcripts if a relevant database is found
Time Frame: By December 2023
Access Criteria: Dependent on the database chosen

REFERENCES:
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Bartlett YK, Farmer A, Rea R, French DP. Use of Brief Messages Based on Behavior Change Techniques to Encourage Medication Adherence in People With Type 2 Diabetes: Developmental Studies. J Med Internet Res. 2020 May 13;22(5):e15989. doi: 10.2196/15989. PMID 32401214